CLINICAL TRIAL: NCT04200508
Title: Cluster Randomized Trial With Cross-over of Targeted Gown and Glove Intervention to Prevent Staphylococcus Aureus and Carbapenem-resistant Gram-negative Bacteria Acquisition in Community-based Nursing Homes
Brief Title: Targeted Gown and Glove Intervention in Nursing Homes
Acronym: TAGG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to COVID-19 in March 2022. It will not resume because the intervention, enhanced barrier precautions, has been recommended by the CDC and Prevention for nursing homes and is currently being implemented.
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Mary-Claire Roghmann, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HP-00088648
Record Dates: First submitted 2019-12-06; First posted 2019-12-16 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Staphylococcus Aureus; Carbapenem Resistant Gram Negative Bacteria
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Intervention Model Description: Nursing home units with a mix of long- and short-stay residents will be the unit of analysis. All nursing homes participating will go through a 8-12 week baseline. Two nursing homes will be randomized to perform the intervention, while the other two continue with an extended baseline. After 8-12 weeks, there will be a washout period of 4 weeks and then the nursing homes will crossover; nursing homes that were in the intervention arm will go back to baseline and those in the extended baseline will perform the intervention. Throughout each study period, we will be assessing Staphylococcus aureus and carbapenem resistant gram-negative bacteria acquisition among residents on each of the nursing homes units being studied
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Targeted gown and glove use for high risk care activities in high risk residents
  Interventions: Other: Targeted gown and gloves use
- Baseline (No Intervention): Standard of Care

INTERVENTIONS:
Other: Targeted gown and gloves use — Gown and glove use for high risk care activities in high risk residents
  Arms: Intervention

SUMMARY:
This project will assess the feasibility of a cluster-randomized trial with crossover of our intervention, targeted gown and glove use, among high-risk residents of community nursing homes to prevent Staphylococcus aureus and carbapenem gram negative bacteria acquisition and infection.

DETAILED DESCRIPTION:
Nursing homes are settings with a high rate of Staphylococcus aureus (SA) and carbapenem -resistant Gram-negative bacteria (C-GNB) acquisition, which can lead to infection, particularly for short stay residents who are recovering from an acute illness. The current standard of care for preventing antibiotic-resistant bacteria acquisition in nursing homes is Standard Precautions (gowns and gloves for anticipated contact with blood, body fluids, skin breakdown or mucous membranes) for all residents.

The intervention is gown and glove use for high-risk care of high-risk residents based on prior research showing the increased risk of transmission from residents to healthcare workers' hands and clothing associated with certain care activities. Rather than wearing gowns and gloves for all care activities to prevent transmission (as would be indicated for Contact Precautions), gown and glove use is targeted to specific resident care activities (e.g., bathing, dressing, and toileting) with prolonged resident-staff contact.

The intervention will occur on units with a mix of long stay and short stay residents, within the nursing home with the NH as the unit of analysis. The primary outcome will be SA, both methicillin-resistant Staphylococcus aureus (MRSA), and methicillin susceptible Staphylococcus aureus (MSSA), and C-GNB acquisition as determined by surveillance cultures in short stay residents, which is a more frequent outcome than infection. During an 8-12 week baseline period, SA and C-GNB acquisition will be assessed via culture and use of gown and gloves for high-risk care of high-risk residents shall be assessed at all nursing homes. A 4-week training period shall occur for each of the nursing homes prior to the start of the intervention period where the NH staff shall be trained on the targeted gown and glove approach. The training period shall be followed by an 8-12 week intervention period, during which SA and C-GNB acquisition shall be assessed via culture and use of own and gloves for high risk care of high-risk residents shall again be assessed and compared to the baseline period. Each nursing home shall act as their own control, via direct comparison of each nursing home during the intervention to itself during the baseline period, reducing variability. The two nursing homes in group 1 shall be trained on and then implement the intervention during study period 1, while the two nursing homes in group 2 continue the baseline period. The two nursing homes in group 2 shall then undergo training and implementation the intervention in study period 2 while the group 1 nursing homes have a washout period then the cross-over baseline observations and cultures. The baseline period, intervention period, and the cross-over baseline period shall each continue for 8-12 weeks aiming for at least 100 resident admissions during each of the study periods (baseline period, intervention period, and cross-over baseline period). Some facilities may not reach 100, but the average across must exceed 100 each.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Reside in a participating nursing home

Exclusion Criteria:

* Identified by nursing home staff as combative or with other behavioral problems which could lead to agitation if approached by project staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Staphylococcus aureus acquisition as determined by surveillance cultures in short stay residents | 1 year
  Rate of Staphylococcus aureus acquisition by short stay residents comparing the baseline and intervention periods
Carbapenem-resistant gram-negative bacteria acquisition as determined by surveillance cultures in short stay residents | 1 year
  Rate of carbapenem-resistant gram-negative bacteria acquisition by short stay residents comparing the baseline and intervention periods
Percentage of high risk patients correctly identified and placed on contact precautions | 1 year
  Percentage of high risk patients with wound and medical devices correctly identified and placed on contact precautions
Percentage of healthcare workers using personal protective equipment during high risk care | 1 year
  Percentage of healthcare workers using personal protective equipment when performing high risk care on high-risk residents

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No